CLINICAL TRIAL: NCT02391922
Title: Bedre førstehjelp Med førstehjelpstrening og AMK-veiledning?
Brief Title: Better First Aid With First Aid Training and Dispatcher Central Instructions?
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Could not recruit eligible PhD-candidate to take on the project
Sponsor: University of Tromso (Other)
Collaborators: Norway: Helgeland Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2014/1844(REK)
Record Dates: First submitted 2014-12-31; First posted 2015-03-18 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Injury
Keywords: out of hospital cardiac arrest; first aid
MeSH Terms: conditions — Wounds and Injuries; Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- No first aid course, No dipatch instruction (No Intervention): Participants' first aid skills are tested in two scenarios without prior first aid course and no dispatch instructions during the scenarios
- First aid course, No dispatch instructions (Active Comparator): Participants' first aid skills are tested in two scenarios 4 to 5 months after receiving a first aid course and no dispatch instructions during the scenarios
  Interventions: Behavioral: First aid course
- First aid course, dispatch instructions (Active Comparator): Participants' first aid skills are tested in two scenarios 4 to 5 months after receiving a first aid course and they are given instructions from emergency dispatch by phone during the test scenarios
  Interventions: Behavioral: First aid course; Behavioral: First aid instructions by mobile phone
- No first aid course, dispatch instructions (Active Comparator): Participants' first aid skills are tested in two scenarios without prior first aid course, and they are given instructions from emergency dispatch by phone during the test scenarios
  Interventions: Behavioral: First aid instructions by mobile phone

INTERVENTIONS:
Behavioral: First aid course
  Arms: First aid course, No dispatch instructions; First aid course, dispatch instructions
Behavioral: First aid instructions by mobile phone
  Arms: First aid course, dispatch instructions; No first aid course, dispatch instructions

SUMMARY:
The study evaluates the effect of a first aid course on first aid skills compared to no training. The study also evaluates the effect of first-aid instructions given by emergency dispatch central over mobile phone on first aid performance to no instructions.

Half the participants will perform first aid in two scenarios prior to first aid training. Half the participants will perform first aid in two scenarios 4 to 5 months after attending a first aid course. Half the participants (overall) will receive first aid instructions by mobile phone during the scenarios.

ELIGIBILITY:
Inclusion Criteria:

* Students in high school/college

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2016-06 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
First aid performance after first aid course | 4-5 months
  First aid performance 4-5 months after first aid course. Measured by a combined score from assigning specific first aid measures a score for being performed.
First aid performance during first aid instructions by phone | Baseline
  First aid performance. Measured by a combined score from assigning specific first aid measures a score for being performed.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tromso, Tromsø, Norway